CLINICAL TRIAL: NCT00756795
Title: Increasing Physical Activity of Patients With Head and Neck Cancer (I-PAP Study)
Acronym: I-PAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI chose not to continue with this unfunded study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0053-08-FB
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Attention Control (Experimental): 5ml of blood will be collected from each blood draw at baseline and post-intervention to assay for Interleukin-6 level.
  Patient will be taught how to keep the Activity diary to record walking and physical activities.
  Structured Interview will be conducted at baseline and post-intervention. All patients will receive 3 reminder phone calls during the first week of study and 10 minutes social visits in the following weeks by study coordinator on a weekly basis
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — 5ml of blood will be collected from each blood draw at baseline and post-intervention to assay for Interleukin-6 level.
  Structured Interview will be conducted at baseline and post-intervention.
  Patients assigned to the Intervention group will be given pedometers to obtain distance walked. In addition, patient will be taught how to keep the Exercise diary to record walking and physical activities.
  All patients will receive 3 reminder phone calls during the first week of study and 10 minutes social visits in the following weeks by study coordinator on a weekly basis.
  Other Names: Digi-Walker ™ Pedometer: SW-701

SUMMARY:
Generally, patients who have undergone treatments for Head Neck Cancer have a decreased quality of life and experience depression and fatigue. Regular physical activity improves emotional well-being, increases immunological response, improves wound healing, lessens fatigue and improves general functionality and quality of life.

This study will determine effectiveness of the 12-week exercise intervention program, determine if physically active patients differ in quality of life, depression and fatigue during the course of the study, and determine if the change in physical activity levels is related to changes in immune responses.

DETAILED DESCRIPTION:
The general hypothesis of this research is that patients who have undergone treatments for Head Neck Cancer have a decreased quality of life and experience depression and fatigue. Increasing and sustaining physical activity of these patients will improve their emotional well-beings, increase their immunological response, improve wound healing, lessen fatigue and improve their general functionality and quality of life.

The purposes of this study are to: (1) determine the effectiveness of the 12-week exercise intervention program in increasing physical activity in head and neck cancer patients; (2) determine if physically active patients differ in quality of life, depression and fatigue during the course of the study; and (3) determine if the change in physical activity levels is related to changes in the immune responses in human.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or above (Nebraska legal age).
2. Patients diagnosed with HNC who are seen at the University of Nebraska Medical Center.
3. Patients who have undergone chemotherapy, radiation and/or surgery for their cancer.
4. Patients who have completed their cancer treatment at least 3 months prior.
5. Patients who have consented to participate in this study with approval by their physicians.
6. Patients who have no significant mental impairment.

Exclusion Criteria:

1. Patients who are on enteral feeding.
2. Patients who are not able to walk or whose surgeons report that walking is not advisable.
3. Patients diagnosed with Lymphoma, Thyroid cancer or Melanoma.
4. Patients who are on antidepressant medications.
5. Patients who are unwilling to return to the clinic at the end of the study - after 12 weeks of intervention.
6. Patients participating in another research study involving a therapeutic intervention.
7. Patients with chronic medical and orthopedic conditions that would preclude physical activity (e.g., congestive heart failure, recent knee or hip replacements).
8. Patients who are at 18 months or more after the start of cancer treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2010-08-05 (Actual); Study Completion 2010-08-05 (Actual)

PRIMARY OUTCOMES:
Self-report of physical activity behavior (duration, intensity and frequency) | Baseline and Post Intervention
  Participants will be taught how to keep the Activity diary to record walking and physical activities.

SECONDARY OUTCOMES:
Plasma IL-6 Concentration | Baseline and Post Intervention
  5ml of blood will be collected from each blood draw at baseline and post-intervention to assay for Interleukin-6 level.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin G Wee, Principal Investigator — University of Nebraska